CLINICAL TRIAL: NCT04269460
Title: Comparison of Ultrasound Guided Subcostal Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Pediatrics Undergoing Pyeloplasty.
Brief Title: Ultrasound Guided Subcostal Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Pediatrics Undergoing Pyeloplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, lecturer of anesthesia, Cairo university hospitals, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D-41-2019
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pain Management; Pediatrics; Anesthesia
Keywords: ultrasound; quadratus lumborum; subcostal TAP; pediatrics; pyeloplasty
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subcostal transversus abdominis plane block (sTAP) (Active Comparator): patients will be in the supine position; after preparing the skin with with povidone iodine, a high frequency (5-10 MHz) ultrasound probe will be used tp identify the rectus abdominis muscle, then 1 mL/Kg of bupivacaine 0.25% will be injected in the plane between rectus abdominis and transversus abdominis muscles.The patient will then be positioned for the procedure if other than supine position is chosen.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution [MARCAINE]
- quadratus lumborum block (QLB) (Active Comparator): patients will be positioned in the lateral decubitus position so that the blocked side will be the uppermost one. After skin sterilization with povidone iodine the ultrasound probe will be positioned to identify the quadratus lumborum muscle. then 1 mL/Kg of bupivacaine 0.25% will be injected behind the QL muscle on the lateral border of the erector spinae muscle.The patient will then be positioned for the procedure if other than lateral decubitus position is chosen.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution [MARCAINE]

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.25% Injection Solution [MARCAINE] — preoperative ultrasound guided subcostal TAP block and Quadratus lumborum block using 1 ml/kg of Bupivacaine Hydrochloride 0.25%in pediatric patients undergoing pyeloplasty surgeries.

SUMMARY:
The aim of this work to compare the analgesic efficacy of preoperative ultrasound guided subcostal TAP block and Quadratus lumborum block in pediatric patients undergoing pyeloplasty surgeries.

DETAILED DESCRIPTION:
This randomized, controlled study is designed to:

* Assess the quality of perioperative analgesia (intraoperative hemodynamics, postoperative pain score and analgesic consumption) provided by ultrasound guided subcostal TAP and quadratus lumborum blocks in pediatrics undergoing pyeloplasty surgeries.
* Compare the efficacy and safety of both blocks in pediatrics undergoing pyeloplasty surgery.

Hypothesis

Following approval from research and ethics committee of anesthesia department, Faculty of Medicine, Cairo University, children will be pre-medicated by intramuscular injection of atropine 0.02 mg/Kg, midazolam 0.2 mg/Kg and ketamine 2 mg/ Kg before admission to operation theater (OR).

Upon arrival to OR; continuous electrocardiography (ECG), pulse oximetry, non-invasive arterial blood pressure will be applied and baseline readings will be recorded, then general anesthesia will be induced by 8% sevoflurane and 50% air in oxygen. Peripheral venous cannula will be inserted after loss of consciousness. If a patient had an intravenous (IV) cannula, induction will be performed using 1.5-2.5 mg/kg propofol, in both situations atracurium at a dose of 0.5 mg/kg will be given intravenously to facilitate endotracheal intubation and fentanyl at a dose 2 µg/kg will be given to abolish stress response of intubation. Anesthesia will be maintained by using 1-1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

Patient positioning and preparation for the block:

For the (sTAP) group (n=39): patients will be in the supine position; after preparing the skin with with povidone iodine, a high frequency (5-10 MHz) ultrasound probe will be placed obliquely on the upper abdominal wall, along the surgical site subcostal margin near the midline. After identifying the rectus abdominis muscle, we will gradually move the ultrasound probe laterally along the subcostal margin until we identify the transversus abdominis muscle lying posterior to the rectus muscle. A 22 G echogenic needle using the in-plane technique will be inserted medially near the xiphoid process aiming towards the iliac crest, then 1 mL/Kg of bupivacaine 0.25% will be injected in the plane between rectus abdominis and transversus abdominis muscles. The patient will then be positioned for the procedure if other than supine position is chosen.

For the (QLB) group (n=39): patients will be positioned in the lateral decubitus position so that the blocked side will be the uppermost one. After skin sterilization with povidone iodine the ultrasound probe will be positioned between the iliac crest and the costal margin at the level of the anterior axillary line to identify the three thin parallel muscles of the anterolateral abdominal wall. The probe will be moved posteriorly following the narrowing of the muscles until the muscle fibers of transversus abdominis muscles taper off into its aponeurosis at the level of the posterior axillary line where the quadratus lumborum muscle is identified. The posterior aspect of the QL muscle is confirmed and a 22 G echogenic needle will be inserted using an in-plane technique from anterolateral to posteromedial towards this posterior aspect of the QL muscle. 1 mL/Kg of bupivacaine 0.25% will be injected behind the QL muscle on the lateral border of the erector spinae muscle. The patient will then be positioned for the procedure if other than lateral decubitus position is chosen.

Vital signs (heart rate (HR) and non-invasive blood pressure) will be recorded at the onset of the block then every 15 minutes intraoperatively, and every 4 hours postoperatively for a period of 24 hours. Fentanyl 0.5 µg /kg as rescue analgesia will be given intraoperatively if HR and or systolic BP increased >20% of baseline up to maximum 5 µg/ kg.

After skin closure, inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered IV after return of patient's spontaneous breathing. Patients will then be transferred to post anesthesia care unit (PACU) for 60 min to complete recovery and monitoring.

Postoperative assessment and analgesic regimen:

The Face, Legs, Activity, Cry, Consolability scale (FLACC) (table 1) will be assessed immediately postoperative in the PACU and every 4 hours in the ward for 24 hours. The time to the first request of rescue postoperative analgesic will be: "the time interval between the local anesthesia injection and the first request to postoperative analgesia (patients first complain of pain and or FLACC score ≥4)". an intravenous paracetamol 15mg/kg will be given immediately postoperative and will be repeated every 6 hours. Persistent or breakthrough pain will be managed with incremental intravenous morphine at a dose of 0.05-0.1mg/kg to maintain resting FLACC scale ˂ 4 (maximum dose 0.3mg/kg). Cumulative 24 hours analgesic consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) physical status I-II.
* Age: 3 months to 5 years.
* Undergoing pyeloplasty surgeries.

Exclusion Criteria:

* Refusal of parents.
* Patients with coagulation disorders (INR > 1.5 and/or platelets < 100 000).
* History of allergic reactions to local anesthetics.
* Rash or signs of infection at the injection site.
* Emergency surgery.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score by The Face, Legs, Activity, Cry, Consolability scale (FLACC) scale at 12 hours | 24 hours
  The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
• Time to first request of postoperative rescue analgesics | 24 hours
  the time interval between the local anesthesia injection and the first request to postoperative analgesia (patients first complain of pain and or FLACC score ≥4.
• Total consumption of opioids | 24 hours
• Block performance time | 24 hours
  time from probe contact with skin till needle withdrawal.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided